CLINICAL TRIAL: NCT06670378
Title: A Multicentre, Prospective, Longitudinal and Observational Natural History Study for Patients With Nemaline Myopathy in the United Kingdom: NatHis-NM-MDUK
Brief Title: Natural History Study for Patients With Nemaline Myopathy in the UK
Acronym: NatHis-NM-MDUK
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Muscular Dystrophy UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: NatHis-NM-MDUK; 24/EE/0114 (Other: REC)
Record Dates: First submitted 2024-09-09; First posted 2024-11-01 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-08

CONDITIONS: Nemaline Myopathy
MeSH Terms: conditions — Myopathies, Nemaline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Up to 15mls of blood will be taken and no more than 0.8 ml/kg will be sampled. These samples will be processed to obtain acellular plasma and DNA which will be stored in the MRC Centre for Neuromuscular Diseases (MRC CNMD) Biobank London is based at the UCL Institute of Neurology and the UCL Great Ormond Street Institute of Child Health.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nemaline myopathy patients: Patients of any age and ability with a genetic and clinical diagnosis of Nemaline myopathy with no significant comorbidities. All patients will be evaluated for the natural clinical progression of the disease using scales and questionnaires for the assessment of motor function, breathing, swallow function and Quality of life and fatigue. In addition it will collect data on continuous movement and gait analysis using real world data and wearable sensors (Syde and Maiju), blood samples for future genetic and proteomic analysis and respiratory analysis using ventilatory and thoraco-abdominal pattern for some paediatric participants.

SUMMARY:
The goal of this study is to to learn more about what assessments would be useful to measure for NM and what normally happens during the lives of people with NM to support future clinical trial development.

DETAILED DESCRIPTION:
Current treatments for people living with nemaline myopathy are supportive only. Several potential therapies are in development which may be available in the next 5-10 years. The barrier to these becoming available is that there is little data available on the natural progression (natural history) of nemaline myopathy. This means that it would be difficult to do a clinical trial of a treatment because it is not known which assessments would be useful to measure or what normally happens during the lives of people with NM.This study aims to better define the natural history and disease specific outcome measures and biomarkers.

This study will comprehensively evaluate the natural clinical progression of the disease using medical data and examination findings, scales and questionnaires for the assessment of motor function, breathing, swallow function and Quality of life and fatigue. In addition it will collect data on continuous movement and gait analysis using real world data and wearable sensors (Syde and Maiju), blood samples for future genetic and proteomic analysis and respiratory analysis using ventilatory and thoraco-abdominal pattern for paediatric participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient and/or parent or legal guardian must be willing and have the ability to provide written informed consent for participation in the study.
* Male or Female
* Any age
* Diagnosis of NM which in most cases includes having a disease-causing variant/s in one of the known NM causative genes and a consistent clinical phenotype.

Exclusion Criteria:

* Any confirmed chronic or acute condition or disease affecting any system(s), which could interfere with the results of the study and/or the compliance with the study procedures. This will be subject to the clinical judgement of the Chief Investigator (CI) and/or the Principal Investigator (PI).
* Clinically significant medical finding on the physical examination other than NM that, in the judgment of the Investigator, will make the patient unsuitable for participation in, and/or completion of the study procedures.
* Participants of ongoing (interventional) clinical trials that assess the efficacy of potential treatments will be excluded as assessments need to be done on the basis that represent the natural progression of NM.
* Safety concerns. This includes anything that might put the participant and/or their Parent(s) or Guardian(s) at risk through participating in the study potentially including but not limited to: Safeguarding concerns, Social Issues and Health issues.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Male or Female
  * Any age
  * Diagnosis of NM which in most cases includes having a disease-causing variant/s in one of the known NM causative genes and a consistent clinical phenotype.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
To observe the natural clinical progression of NM in patients not receiving any disease-modifying intervention | Baseline, 6 months (age <18 years only), 12months, 18 months (age <18 years only) 24 months, 36 months.
  Collection of retrospective and prospective clinical data at baseline visit
To observe the natural clinical progression of NM in patients not receiving any disease-modifying intervention | Baseline, 6 months (age <18 years only), 12months, 18 months (age <18 years only) 24 months, 36 months.
  Standard Medical and Neurological examination
To observe the natural clinical progression of NM in patients not receiving any disease-modifying intervention | Baseline, 6 months (age <18 years only), 12months, 18 months (age <18 years only) 24 months, 36 months.
  Questionnaires focusing on quality of life:
  All ages = PROMIS - 29 profile v2.1
To observe the natural clinical progression of NM in patients not receiving any disease-modifying intervention | Baseline, 6 months (age <18 years only), 12months, 18 months (age <18 years only) 24 months, 36 months.
  Physio assessment for motor outcome measures and assessment is depend on age:
  0-1 years old (dependent on ability) CHOP-INTEND, HINE2, Peabody and MFM32
  2-4 years (dependent on ability) MFM32, NSAD, Peabody
  5 and over (dependent on ability) MFM32, NSAD, PUL, Myogrip, myopinch, 4SCT, 6MWY, 100mWRT
To observe the natural clinical progression of NM in patients not receiving any disease-modifying intervention | Baseline, 6 months (age <18 years only), 12months, 18 months (age <18 years only) 24 months, 36 months.
  Respiratory outcome measured dependent on age 0-1 years old (dependent on ability) Time on/off ventilator
  2-4 years (dependent on ability) Time on/off ventilator, SNIP
  5 and over (dependent on ability) Time on/off ventilator, Spirometry, MIP/MEP, SNIP

SECONDARY OUTCOMES:
To quantify the health economic burden of nemaline myopathy | Baseline, 12months, 24 months, 36 months.
  Health Utilities Index 3 (HUI3)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Laurent Servais, Study Chair — MDUK Oxford Neuromuscular Centre, University of Oxford
Locations (4):
- United Kingdom (4):
  - Department of Paediatric Neurology - Neuromuscular Service, Evelina Children's Hospital, London
  - Dubowitz Neuromuscular Centre, UCL Great Ormond Street Hospital, London
  - John Walton Muscular Dystrophy Research Centre, Newcastle University, Newcastle
  - MDUK Oxford Neuromuscular Centre, University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: Undecided